CLINICAL TRIAL: NCT00984906
Title: Inspiratory Flow Parameters and Device Handling With Empty Device-metered Dry Powder Inhalers, Easyhaler and Turbuhaler; an Open, Randomised, Multi Centre Study in Patients With Asthma or COPD
Brief Title: Inspiratory Flow Parameters and Handling of Easyhaler and Turbuhaler Inhalers
Acronym: PIFECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Satu Lähelmä/Clinical Study Director, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3103003
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Empty Easyhaler type A (Other)
  Interventions: Other: Empty inhalers
- Empty Easyhaler type B (Other)
  Interventions: Other: Empty inhalers
- Empty Turbohaler (Other)
  Interventions: Other: Empty inhalers

INTERVENTIONS:
Other: Empty inhalers — Empty Easyhaler inhalers (type A and type B) and empty Turbohaler inhaler
  Other Names: Empty device-metered dry powder inhaler Easyhaler (type A); Empty device-metered dry powder inhaler Easyhaler (type B); Empty device-metered dry powder inhaler Turbohaler

SUMMARY:
The aim of the study is to measure the inspiratory flow that the different patient groups (asthmatic children, adults and elderly, as well as chronic obstructive pulmonary disease (COPD) patients) generate through empty Easyhaler (two versions) and Turbuhaler inhalers. In addition, the handling and acceptability of the inhalers will be compared in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Documented diagnosis of asthma and/or COPD (a range of different severities for both diseases).
* Age: 6 years or above.

Exclusion Criteria:

* Any severe chronic respiratory disease other than asthma or COPD.
* Acute respiratory infection.
* Concurrent participation in a clinical drug study.
* Inability to perform repeatable spirometric measurements.
* Any medical condition that in the opinion of the investigator would endanger the subject if he/she participates in the study (such as contraindications to spirometry).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Peak inspiratory flow rate through the empty Easyhaler and Turbohaler inhalers | 1 Day

SECONDARY OUTCOMES:
Other inspiratory flow parameters through the empty Easyhaler and Turbohaler inhalers measured at the same time with the peak inspiratory flow rate. | 1 Day
Handling of the devices in the subpopulation of asthmatic children | 1 Day
Acceptability of the inhalers in the subpopulation of asthmatic children | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Satu Lähelmä, M.Sc.(Pharm), Study Director — Orion Corporation, Orion Pharma
Locations (4):
- Finland (2):
  - Jorvi hospital, Helsinki
  - Skin and Allergy hospital, Helsinki
- United Kingdom (2):
  - Northern General Hospital, Sheffield
  - Sheffield Children's Hospital, Sheffield